CLINICAL TRIAL: NCT03176953
Title: Combining Topiramate and Prolonged Exposure for PTSD and Alcohol Use Disorder
Brief Title: Topiramate and Prolonged Exposure
Acronym: TOP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2412-R
Record Dates: First submitted 2017-05-30; First posted 2017-06-06 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: PTSD and Alcohol Use Disorder
Keywords: PTSD; alcohol use disorder; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of two conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study. Only pharmacist will have access to randomization table.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- prolonged exposure + topiramate (Experimental): psychotherapy plus active medication
  Interventions: Drug: topiramate; Behavioral: prolonged exposure
- prolonged exposure + placebo (Active Comparator): psychotherapy plus placebo medication
  Interventions: Behavioral: prolonged exposure; Drug: placebo

INTERVENTIONS:
Drug: topiramate — active medication
  Arms: prolonged exposure + topiramate
Behavioral: prolonged exposure — psychotherapy
Drug: placebo — non-active medication
  Arms: prolonged exposure + placebo

SUMMARY:
Alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) frequently co-occur, and having both disorders is associated with greater psychological and functional impairment than having either disorder alone. The most effective PTSD treatment, prolonged exposure (PE) is sometimes less effective when individuals also have AUD. Anti-relapse medication appears promising to improve the effectiveness of PE to help individuals reduce alcohol use and PTSD symptoms and improve functioning. This study compares PE with and without topiramate, a medication shown to both reduce drinking and PTSD symptoms, with the hypothesis that combined PE and topiramate will be more effective than PE and placebo. The aim of this grant is to improve treatment outcomes for Veterans with AUD and PTSD.

DETAILED DESCRIPTION:
Objectives. Alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) frequently co-occur, and having one condition worsens the course of the other. Individuals with both disorders exhibit worse functioning across a number of domains than individuals with either disorder alone. Prolonged exposure therapy (PE) is among the most effective treatments for PTSD. PE has been rated as a frontline treatment by multiple guidelines and reviews including the VA/DoD Clinical Practice Guidelines for the treatment of PTSD. However, in studies of individuals with PTSD and AUD, changes in alcohol use are only slightly better than in control or standard care conditions, reductions in PTSD symptoms are sometimes modest relative to studies of PE in PTSD patients without AUD, and rates of drop out from treatment are high. Combining PE with medication to curb drinking shows promise to improve upon the effectiveness of PE for individuals with comorbid AUD and PTSD, although thus far few studies have examined combining psychotherapy and medication. Topiramate is the single medication that has shown effectiveness for both AUD and PTSD and shows promise for reducing drinking among individuals with AUD and PTSD. However, the effect of adding topiramate to PE to treat comorbid AUD/PTSD has yet to be examined. The critical next step is to test a best practice PTSD treatment, PE, together with a promising pharmacological agent, topiramate, which has been found to be effective for both AUD and PTSD. Innovation: This application seeks to shift current clinical practice paradigms. A refinement to existing interventions is proposed through integration of two evidence based treatments.

Methodology. The investigators propose to use a randomized, controlled, double blind study design to examine the effect of adding topiramate (TOP) to a best practice treatment for PTSD, PE. Participants will be 120 male and female Veterans from all services with AUD and PTSD. The investigators' primary aims are to determine the relative efficacy of PE+topiramate, as compared to PE+placebo, in reducing problematic drinking, reducing PTSD symptoms, and improving functioning and quality of life among Veterans with comorbid AUD/PTSD at post-treatment and 3- and 6-month post-treatment follow-up. The investigators will explore the extent to which decreases in drinking and PTSD symptoms lead to improvement in functioning.

The proposed study has the potential to improve functional and psychological recovery for a highly prevalent and highly impaired population of Veterans. This study will test a novel and innovative combination of psychotherapy and medication with the goal of improving the care of Veterans. The successful completion of this project will help change the practices that drive treatment for Veterans who have both AUD and PTSD. The fundamental rationale for this study is to improve the evidence base that informs how patients with AUD and PTSD can attain sustained recovery from both of these disorders. The investigators will also explore whether changes in PTSD symptoms in the PE+TOP condition are partially explained by reductions in alcohol cravings.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans of the U.S. military and/or Reserve/National Guard members,
2. at least 18 years of age,
3. survivors of a psychological trauma meeting DSM-5 criterion A, and are at least one month post-trauma,
4. have current DSM-5 diagnoses of AUD and PTSD based on semi-structured diagnostic interviews,
5. have at least 20 days of heavy drinking (>= 5 drinks/day for men and >= 4/drinks per day for women) in the last 90 days spent in a non-restricted environment and meet criteria for heavy drinking at least 4 days in the last 30 days prior to screening,
6. are not currently receiving trauma-focused psychotherapy,
7. are literate in English and intend to stay in the San Diego area during the study,
8. are willing to attend psychotherapy, medication, and assessment sessions,
9. trying or planning to try to cut down on or abstain from alcohol,
10. for females of childbearing potential, agree to use an approved form of contraception for the duration of the study, including hormonal contraceptives (e.g., oral contraceptives or implantable devices), intrauterine device (IUD), or double barrier methods (e.g., diaphragm with spermicidal condom); barrier method is preferred as topiramate may make birth control less effective,
11. Individuals with clinically significant renal disease and/or impaired renal function, as defined by clinically significant elevation of blood urea nitrogen (BUN) or creatinine or an estimated creatinine clearance of < 60 mL/min, can be included with physician approval, however the dosing schedule and maximum dose will be adjusted in accordance with FDA prescribing guidelines,
12. if individual is on another addiction medication, they should be on a stable approved addiction medication dose (at least two weeks before starting study drug) throughout the study,
13. are capable of giving informed consent.

Exclusion Criteria:

1. Subjects known to have clinically significant unstable medical or psychiatric conditions, where participation is deemed by investigators and study physicians to be risky, including but not limited to:

   * AST and/or ALT >5 times the upper limit of the normal range and/or an increased serum bilirubin >2 times the upper limit of normal.
   * Seizure disorders
2. have been treated with Topiramate for any reason in the past and discontinued the drug due to hypersensitivity reaction
3. in the opinion of the investigator, should not be enrolled because of the precautions, warnings, or contraindications listed on the Topiramate package insert, (e.g., certain types of glaucoma),
4. are pregnant, lactating, or plan to become pregnant during the period of participation in the study
5. in the judgment of the investigator, represent a significant risk of suicidal or homicidal behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya B. Norman, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolonged Exposure + Topiramate | Prolonged Exposure + Placebo
Started | 50 | 50
Completed | 41 | 40
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Population: randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure + Topiramate | Prolonged Exposure + Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.86 (12.39) | 44.67 (12.90) | 45.27 (12.60)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  sex: male | 42 | 42 | 84
  sex: female | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 36 | 32 | 68
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 15 | 22
  White | 33 | 28 | 61
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Education [Count of Participants; unit: Participants]
  GED/High School Diploma | 7 | 7 | 14
  Some college | 23 | 22 | 45
  College degree | 15 | 17 | 32
  Missing | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: CAPS-5 Change
Description: PTSD symptom diagnostic interview CAPS-5 score range = 0 - 80 Higher scores = more severe PTSD symptoms
Time Frame: Change from baseline to 16 weeks
Population: All randomized participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prolonged Exposure + Topiramate | Prolonged Exposure + Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  baseline CAPS | 36.720 (1.794) | 38.600 (1.794)
  16-week CAPS | 21.006 (1.988) | 29.872 (2.016)

2. Primary Outcome: Timeline Followback Interview (TLFB)
Description: substance use severity score range = 0 - 100% of heavy drinking days higher scores = greater percentage of total days that included heavy drinking
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Prolonged Exposure + Topiramate | Prolonged Exposure + Placebo
Number analyzed (Participants) | 50 | 50
percentage of days
  Baseline | 53.5 (3.6) | 52.1 (3.6)
  16 week | 10.8 (4.1) | 16.2 (4.2)

ADVERSE EVENTS:
Time Frame: Duration of study participation - 10 months
Description: Definitions did not differ. Systematic assessment by clinicians during treatment phase and assessors during follow-up phase.
Arm/Group | Prolonged Exposure + Topiramate | Prolonged Exposure + Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 4/50 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure + Topiramate (N=50) | Prolonged Exposure + Placebo (N=50)
psychiatric hospitalization (Psychiatric disorders) | 2 (2) | 0 (0)
arrest (Social circumstances) | 1 (1) | 1 (1)
severe headache (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure + Topiramate (N=50) | Prolonged Exposure + Placebo (N=50)
acidosis (Endocrine disorders) | 1 (1) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
physical injury due to fighting or non-suicidal self-harm (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
incarceration due to parole violation (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03176953/Prot_SAP_000.pdf